CLINICAL TRIAL: NCT06764966
Title: A Pilot Study of Statin and Beta Blocker Use in Patients with Decompensated Cirrhosis
Brief Title: Statin and Beta Blocker Use in Patients with Decompensated Cirrhosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Nadeem Anwar, Section Chair, Gastroenterology, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-1117
Record Dates: First submitted 2025-01-07; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Decompensated Liver Cirrhosis; Cirrhosis; Decompensated Cirrhosis of Liver; Decompensated Cirrhosis and Ascites
Keywords: Decompensated Cirrhosis; Decompensated Liver Disease; Statins; Beta-Blockers; Cirrhosis
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NSBB plus statin (Active Comparator): Atorvastatin 20 mg once daily along with previously prescribed NSBB
  Interventions: Drug: Atorvastatin 20 mg
- NSBB plus placebo (Placebo Comparator): Placebo once daily along with previously prescribed NSBB
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin 20 mg — Atorvastatin 20 mg Once Daily with previously prescribed Non Selective Beta-Blocker
  Arms: NSBB plus statin
Drug: Placebo — Placebo Once Daily along with previously prescribed Non Selective Beta Blocker
  Arms: NSBB plus placebo

SUMMARY:
Decompensated cirrhosis (liver disease) occurs when liver function decreases to the extent that serious complications develop and can include internal bleeding, fluid buildup in the abdomen, or mental confusion. This reduced decreased liver function subsequently decreases life expectancy. There is a critical need for strategies to delay progression to decompensation and reduce the occurrence of serious complications. Currently, limited therapeutic options are available for managing decompensated liver disease, with beta-blockers (BB) being the only proven medication with significant benefits in preventing disease progression. Statins have been historically under- prescribed in cirrhosis due to concerns of liver damage. However, there is emerging evidence that statin use may be beneficial and able to lessen liver disease worsening, with studies demonstrating its safety. Thus, we aim to conduct a pilot randomized controlled trial (RCT) study of 50 subjects comparing the outcomes of decompensated cirrhotic patients receiving the statin, atorvastatin, and a non-selective beta-blocker (NSBB) versus those receiving NSBB plus placebo. Both groups will be followed for 12 months to investigate the feasibility, safety, and efficacy of combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients age of 18 years or older diagnosed with any form of decompensated liver disease defined as ascites, hepatic encephalopathy, or variceal bleed presenting at Charleston Area Medical Center (CAMC) Memorial Hospital or CAMC-Gastroenterology Liver Clinic
* Currently on an non-selective beta-blockers agreeing to have their liver disease managed by CAMC-Gastroenterology Liver Clinic as an outpatient for the 12-month follow-up period.

Exclusion Criteria:

* Any patient <18 years of age
* Patients with hepatocellular carcinoma
* Patients with ongoing alcohol use (self-reported consumption of more than one alcoholic drink per week)
* Patients exhibiting high-risk behaviors that could put them at risk for complications including IV substance use and history of medication non-adherence
* Patients currently on statin therapy
* Patients with a history of statin intolerance
* Patients on the waitlist for liver transplantation
* Patients taking medications with known drug interactions with statins
* Patients not able to give informed consent or patients belonging to vulnerable categories as the Federal Regulations or Common Rule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility- compare the number of participants who discontinued study medication for any reason during the 12-month follow-up period | 12 months
Feasibility- compare the number of participants compliant with study treatment | 12 months
  Participants will be considered compliant if they attend four follow-up visits and consume ≥ 75% of study medication (determined by pill counts)

SECONDARY OUTCOMES:
Safety - Adverse events | 12 months
  Rate of reported treatment-related adverse events (muscle pain, muscle injury, liver injury, kidney dysfunction, other)
New Decompensating events | 12 months
  Rate of new decompensating events (ascites, vatical bleeding, worsening jaundice, or encephalopathy) in each arm, time for development of new decompensating event
Hepatic transaminases levels | 12 months
  Number of participants with increases in transaminases by more than five times the upper limit of normal
Survival rate | 12 months
  Rate of survival between the two treatment arms
Transplant-free survival rate | 12 months
  Number of participants without liver transplant during study participation
Rate of Hepatocellular Carcinoma Diagnosis | 12 months
  Number of participants developing Hepatocellular Carcinoma over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Anwar, MD, Principal Investigator — CAMC Health System
Locations (1):
- Charleston Area Medical Center, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No